CLINICAL TRIAL: NCT05061459
Title: The Expression of circANKRD36 as a New Biomarker of Diabetic Nephropathy in Patients With Type 2 Diabetes Mellitus
Brief Title: The Expression of circANKRD36 as a New Biomarker of Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Magdy Hamed Mohamed, Doctor, Assiut University
Other Study IDs: The expression of circANKRD36
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1:: 28 control
  Interventions: Genetic: circANKRD36 as a new biomarker
- Group 2:: 68 T2DM patients
  Interventions: Genetic: circANKRD36 as a new biomarker

INTERVENTIONS:
Genetic: circANKRD36 as a new biomarker — expression levels of circANKRD36 in the development and progression of DN

SUMMARY:
1. To evaluate expression levels of circANKRD36 in the development and progression of DN.
2. To investigate correlation between expression levels of circANKRD36 and stages of DN.
3. To investigate correlation between expression levels of circANKRD36 and pro-inflammatory cytokine (TNF-α and IL-6) in T2DM patients with CKD.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) is one of the most common metabolic disorders that's become a global health burden affecting 463 million people worldwide according to the International Diabetes Federation (IDF). Diabetic nephropathy(DN) is one of the most common secondary complications of DM and is becoming a major cause of morbidity and mortality among diabetic patients . DN is a microvascular complication occurring in approximately 20-40% of patients with T2DM . DN has been described as a glomerular disorder with the following phases: glomerular hyperfiltration, incipient nephropathy, microalbuminuria, overt proteinuria and end-stage renal disorder. Microalbuminuria is the gold standard for the early diagnosis of DN. However, many studies have suggested that it is inadequate and has some drawbacks. Recent novel biomarkers have been accepted for early diagnosis and progression of DN in patients with T2DM . Renal cells are capable of synthesizing pro-inflammatory cytokines such as tumor necrotic factor-alpha (TNF-α), interleukin-1β (IL-1β) and interleukin-6 (IL-6), these cytokines acting in a paracrine or autocrine manner that leading to the development and progression of several renal disorders .Circular RNAs are class of endogenous non coding RNAs and are associated with numerous diseases like T2DM. Circular ankyrin repeat domain 36 (circANKRD36) involved in T2DM and inflammation-associated pathways via interaction with miRNAs, including hsa-miR-3614-3p, hsa-miR-498, and hsa-miR-501-5p. The expression of circANKRD36 was upregulated in peripheral blood leucocytes and was correlated with chronic inflammation in T2DM. Therefore, circANKRD36 can be used as a potential biomarker for screening chronic inflammation in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as Type 2 Diabetes Mellitus

Exclusion Criteria:

* Any other clinically systemic acute or chronic inflammation disease/s.
* Autoimmune disease.
* Any endocrine disease other than T2DM.
* Cancer.
* Chronic hepatic or renal failure.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include 96 (68 patients diagnosed as T2DM and 28 apparently healthy subjects as control group).
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Expression levels of circANKRD36 in the development and progression of DN. | baseline
  circANKRD36 by reverse transcription-quantitative polymerase chain reaction (RT-qPCR)

SECONDARY OUTCOMES:
Correlation between expression levels of circANKRD36 and pro-inflammatory cytokine (TNF-α and IL-6) in the development and progression of DN. | baseline
  pro-inflammatory cytokine TNF-α by enzyme-linked immunosorbent assay (ELISA). IL-6 by Chemiluminescence on Advia centaur XPT.